CLINICAL TRIAL: NCT01145352
Title: Enbrel-JIA Use Results Survey [All-Case Surveillance]
Brief Title: Enbrel-Juvenile Idiopathic Arthritis (JIA) Use Results Survey [All-Case Surveillance]
Acronym: Enbrel-JIA
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0881Y1-4689; B1801130
Record Dates: First submitted 2010-06-09; First posted 2010-06-16 (Estimated); Results first posted 2014-09-04 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-08

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Enbrel-JIA
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Etanercept

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Etanercept (genetical recombination): All patients who administrated ENBREL for active polyarticular juvenile idiopathic arthritis during registered period (2.5 year).
  Interventions: Drug: Etanercept (genetical recombination)

INTERVENTIONS:
Drug: Etanercept (genetical recombination) — All patients who administrated ENBREL for active polyarticular juvenile idiopathic arthritis (restricted to the case of lack of effect by other treatment) during registered period (2.5 year).
  Other Names: Enbrel

SUMMARY:
This surveillance is conducted to survey the followings under the post marketed drug utilization on the patients who are administrated ENBREL as a treatment for active polyarticular JIA.

1. Primary Occurrence status of Adverse Events; incidence of all adverse events, serious adverse events
2. Secondary Factors affecting safety and to confirm the efficacy such as DAS28.

DETAILED DESCRIPTION:
All patients who administrated ENBREL for active polyarticular juvenile idiopathic arthritis during registered period (2.5 year).

ELIGIBILITY:
Inclusion Criteria:

* Patients in active polyarticular JIA (restricted to the case of lack of effect by other treatment) during enrollment period (2.5years).
* Patients receiving Enbrel for JIA as diagnosed by a qualified physician.
* Age 5 - 16 years

Exclusion Criteria:

* Patients not administered ENBREL

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients who administrated ENBREL for active polyarticular juvenile idiopathic arthritis (restricted to the case of lack of effect by other treatment) during registered period (2.5 year).
Sampling Method: Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2009-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Yokohama City University School of, Tokyo, Japan, Japan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881Y1-4689&StudyName=Enbrel-Juvenile%20Idiopathic%20Arthritis%20%28JIA%29%20Use%20Results%20Survey%20%5BAll-Case%20surveillance%5D

RESULTS

PARTICIPANT FLOW:
Groups:
- Etanercept (Genetical Recombination): Participants with polyarticular juvenile idiopathic arthritis (JIA) who received 10 mg or 25 mg lyophilized etanercept (genetical recombination) for subcutaneous injection.
Period: Overall Study
Arm/Group | Etanercept (Genetical Recombination)
Started | 113
Completed | 102
Not Completed | 11
Not completed — Found to have been registered twice | 6
Not completed — Treated before marketing approval | 4
Not completed — Syringe formulation was used | 1

BASELINE CHARACTERISTICS:
Arm/Group | Etanercept (Genetical Recombination)
Number analyzed (Participants) | 102
Age, Customized [Number; unit: participants]
  <5 years | 1
  >= 5 to < 10 years | 24
  >= 10 to < 15 years | 37
  >= 15 to < 20 years | 30
  >= 20 to < 30 years | 10
  >=30 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Related Adverse Events of Etanercept
Description: Adverse events are all unfavorable events, including clinically problematic abnormal changes in laboratory test values, which develop in participants after the administration of Etanercept, irrespective of causal relationship to Etanercept. The causal relationship between an adverse event and Etanercept was evaluated by the sponsor.
Time Frame: 24 weeks
Population: The safety analysis population consisted of the participants who received 10 mg or 25 mg lyophilized etanercept (genetical recombination) for subcutaneous injection indicated for polyarticular JIA after the marketing authorization had been granted.
Measure: Number; unit: participants
Arm/Group | Etanercept (Genetical Recombination)
Number analyzed (Participants) | 102
participants | 22

2. Primary Outcome: Number of Participants With Serious Treatment-Related Adverse Events of Etanercept
Description: Serious treatment-related adverse events are defined as any events that lead to death, life-thretening, hospitalization or prolonged hospitalization, a permanent or remarkable disorder/dysfunction, congenital anormaly/congenital deficiency, or other medically significant events or disorder.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Etanercept (Genetical Recombination)
Number analyzed (Participants) | 102
participants | 1

3. Primary Outcome: Number of Unlisted Treatment-Related Adverse Events of Etanercept
Description: Adverse events are all unfavorable events, including clinically problematic abnormal changes in laboratory test values, which develop in participants after the administration of Etanercept, irrespective of causal relationship to Etanercept. The causal relationship between an adverse event and Etanercept was evaluated by the sponsor. Unlisted treatment-related adverse events were confirmed with listed adverse drug reactions specified in Japanese package insert.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | Etanercept (Genetical Recombination)
Number analyzed (Participants) | 102
events | 3

4. Primary Outcome: Percentage of Good Responders and Moderate Responders Among Participants With European League Against Rheumatism (EULAR) Response Based on DAS28
Description: The Disease Activity Score Based on 28-joints Count based (DAS28-based) EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders: change from baseline >1.2 with DAS28 =< 3.2; moderate responders: change from baseline >1.2 with DAS28 >3.2 or change from baseline >0.6 to =<1.2 with DAS28 =<5.1; non-responders: change from baseline =< 0.6 or change from baseline >0.6 and =<1.2 with DAS28 >5.1.
Time Frame: 24 weeks
Population: The efficacy analysis population consisted of the participants in whom DAS28 (4/ESR) was calculated (N = number of participants evaluated). The last observation carried forward (LOCF) method was used to impute missing data.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept (Genetical Recombination)
Number analyzed (Participants) | 87
Percentage of participants
  At 4 weeks (N = 25) | 72.00 [50.61 to 87.93]
  At 8 weeks (N = 30) | 73.33 [54.11 to 87.72]
  At 12 weeks (N = 31) | 70.97 [51.96 to 85.78]
  At 16 weeks (N = 32) | 75.00 [56.60 to 88.54]
  At 20 weeks (N = 34) | 73.53 [55.64 to 87.12]
  At 24 weeks (N = 46) | 63.04 [47.55 to 76.79]

5. Secondary Outcome: Percentage of Participants With Overall Improvement On Physician's Assessment.
Description: Percentage of participants in whom the efficacy of etanercept was assessed as either markedly effective or effective.
Time Frame: 24 weeks
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Etanercept (Genetical Recombination)
Number analyzed (Participants) | 87
percent
  At 4 weeks (N = 51) | 94.12 [83.76 to 98.77]
  At 8 weeks (N = 63) | 93.65 [84.53 to 98.24]
  At 12 weeks (N = 64) | 93.75 [84.76 to 98.27]
  At 16 weeks (N = 65) | 93.85 [84.99 to 98.30]
  At 20 weeks (N = 67) | 91.04 [81.52 to 96.64]
  At 24 weeks (N = 83) | 95.18 [88.12 to 98.67]

ADVERSE EVENTS:
Description: The frequency of treatment related adverse events during the study
Arm/Group | Etanercept (Genetical Recombination)
Serious Adverse Events (participants affected / at risk) | 1/102
Other Adverse Events (participants affected / at risk) | 27/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etanercept (Genetical Recombination) (N=102)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etanercept (Genetical Recombination) (N=102)
Erythema infectiosum (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 5 (5)
Nasopharyngitis (Infections and infestations) | 4 (4)
Paronychia (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2)
Seasonal allergy (Immune system disorders) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Iritis (Eye disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Injection site erythema (General disorders) | 1 (1)
Injection site reaction (General disorders) | 5 (5)
Malaise (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Alanine aminotransferase increased (Investigations) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1)
Blood beta-D-glucan increased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.